CLINICAL TRIAL: NCT01868334
Title: A Vaccination SOP Toolkit in Diverse Practices Implemented & Tested With RE-AIM
Brief Title: SOP Toolkit in Diverse Practices Implemented & Tested With RE-AIM
Acronym: SOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Richard Zimmerman MD, Principal Investigator, Professor, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CDC-1U01IP000662-01
Record Dates: First submitted 2013-03-20; First posted 2013-06-04 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Adult Influenza Vaccinations; Adult PPSV Vaccinations; Adult Tdap/Td Vaccinations
Keywords: influenza vaccine; PPSV; Tdap; vaccination; adult
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention with the Toolkit (Experimental): Pillar 1: Convenient Vaccination Services Pillar 2: Patient notification Pillar 3: Enhanced Office Systems Pillar 4: Motivation
  13 clinical practices (intervention sites) will receive the Toolkit in Year 1 to increase their adult influenza, PPSV, Tdap/Td vaccination rates. In Year 2, those who choose to continue will "maintain" use of the Toolkit and online resources available but will receive no active intervention from study staff.
  Interventions: Behavioral: Pillar 1: Convenient Vaccination Services; Behavioral: Pillar 2: Patient notification; Behavioral: Pillar 3: Enhanced Office Systems; Behavioral: Pillar 4: Motivation
- 12 clinical practices (control sites) (No Intervention): 12 diverse clinical practices will receive no additional assistance in Year 1 to increase their adult influenza, PPSV, Tdap/Td vaccination rates, they will follow guidelines for usual care. In Year 2 however they will become intervention sites and receive the 4 Pillars Toolkit for use in increasing vaccination rates

INTERVENTIONS:
Behavioral: Pillar 1: Convenient Vaccination Services — Extend Vaccination Season: Begin vaccinating for influenza as soon as vaccine arrives; use every visit as opportunity to vaccinate; extend the season for influenza by vaccinating in January and beyond.
  Use Express Vaccination services such as influenza vaccination clinics, Open access vaccine scheduling (for all vaccines), or dedicated vaccination station. When giving influenza vaccination, screen for need for PPSV/Tdap.
  Arms: Intervention with the Toolkit
Behavioral: Pillar 2: Patient notification — Patient Education: notifying patients of doctor recommendations for vaccination; providing information on express vaccination services via email, autodialer, "on-hold" messages, clinic websites, and/or social media
  Arms: Intervention with the Toolkit
Behavioral: Pillar 3: Enhanced Office Systems — Routine assessment for office systems flow to ensure staff consistently promoting vaccination: utilization of EMR prompts, review of Immunization tabs within EMR, and/or checking vaccination status as part of vital signs when rooming. Empower staff to vaccinate by use of a standing orders program (SOP). Order a sufficient supply of vaccination to cover increased rates
  Arms: Intervention with the Toolkit
Behavioral: Pillar 4: Motivation — Utilization of an Office Immunization Champion who will track overall progress towards their goal - setting a goal of increased rates of 20 to 25% for influenza vaccine; monitoring and sharing progress with staff regularly; and changing office systems flow as needed to increased vaccination rates.
  Arms: Intervention with the Toolkit

SUMMARY:
The purpose of this study is to test whether or not the 4 Pillars Toolkit increases adult Influenza, pneumococcal polysaccharide vaccine (PPSV), tetanus, adult diphtheria and acellular pertussis vaccine (Tdap/Td) vaccination rates. The vaccines are all FDA licensed vaccines and to be used according to national guidelines. The investigators will conduct a randomized cluster trial of this toolkit in diverse primary care practice with electronic medical records (EMRs).

DETAILED DESCRIPTION:
This intervention is a two-region, two-year, stratified randomized cluster trial in 24 primary care practices with EMRs. These practices will be randomly assigned to be intervention or control sites to test this 4 Pillars Toolkit intervention package of evidence-based techniques tailored to their practice structure and culture; one set of practices randomized to intervention in year 1 and the other to control. In year 2, the other set of practices will receive the intervention and community controls may be sought.

These diverse practices consist of: 18 diverse practices from UPMC in western Pennsylvania and 6 diverse practices from large community health centers in a PBRN in Texas.

ELIGIBILITY:
Practice staff and adults in enrolled clinical sites

Inclusion Criteria:

Site inclusion criteria:

* 1) an appropriate adult population: e.g., adults aged 50 years and older;
* 2) currently using an EMR that has prompt ability, such as EpicCare;
* 3) having and keeping immunization data within this EMR

Patient-level inclusion criteria:

* 1) Adults (18 years and above) who are active patients of the enrolled practices (e.g., active patients are those with a visit within the last 12 months)
* 2) All unvaccinated adults without a contraindication are eligible to receive Td/Tdap and influenza, regardless of age and at age 65 years or older are eligible for PPSV.

Exclusion Criteria:

Site exclusion criteria:

* 1) consistent SOP use for the 3 vaccines being studied or high vaccination rates (e.g., 80%)

Patient-level exclusion criteria:

* 1) those with a true contraindication, following the CDC's Guide to Contraindications (attached with the US Recommended Adult Immunization Schedule), such as prior vaccine anaphylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70549 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Patricia Nowalk, PhD, RD, Study Director — University of Pittsburgh, School of Medicine, Department of Family Medicine; Anthony E Brown, MD MPH, Study Director — Baylor College of Medicine
Locations (2):
- United States (2):
  - University of Pittsburgh, School of Medicine, Department of Family Medicine, Pittsburgh, Pennsylvania
  - Baylor Colllege of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lin CJ, Nowalk MP, Pavlik VN, Brown AE, Zhang S, Raviotta JM, Moehling KK, Hawk M, Ricci EM, Middleton DB, Patel S, South-Paul JE, Zimmerman RK. Using the 4 pillars practice transformation program to increase adult influenza vaccination and reduce missed opportunities in a randomized cluster trial. BMC Infect Dis. 2016 Nov 3;16(1):623. doi: 10.1186/s12879-016-1940-1. PMID 27809793
- [Result] Zimmerman RK, Brown AE, Pavlik VN, Moehling KK, Raviotta JM, Lin CJ, Zhang S, Hawk M, Kyle S, Patel S, Ahmed F, Nowalk MP. Using the 4 Pillars Practice Transformation Program to Increase Pneumococcal Immunizations for Older Adults: A Cluster-Randomized Trial. J Am Geriatr Soc. 2017 Jan;65(1):114-122. doi: 10.1111/jgs.14451. Epub 2016 Oct 18. PMID 27755655
- [Result] Nowalk MP, Lin CJ, Pavlik VN, Brown AE, Zhang S, Moehling KK, Raviotta JM, South-Paul JE, Hawk M, Ricci EM, Middleton DB, Patel SA, Ahmed F, Zimmerman RK. Using the 4 Pillars Practice Transformation Program to increase adult Tdap immunization in a randomized controlled cluster trial. Vaccine. 2016 Sep 22;34(41):5026-5033. doi: 10.1016/j.vaccine.2016.07.053. Epub 2016 Aug 26. PMID 27576073

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: clinical practices
Groups:
- Pittsburgh Intervention Sites: Practices: Clinical practices were stratified by metropolitan area (e.g., Pittsburgh) and then randomized into the intervention or control arms within strata.
  Patients: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 6/1/2012 to 5/31/2013 (Tdap, PCV) and 8/1/2012 to 1/31/2013 (influenza), Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Year 1 RCCT Study: Intervention sites were Pittsburgh practices who actively utilized the 4 Pillars Practice Transformation Program during Year 1 to promote increases in adult vaccination rates (N=10).
  Year 2 Pre-post study: Year 2 Pittsburgh practices were control sites from Year 1 (N=8) who now were actively engaged in the intervention and Year 1 sites who continued active use of the intervention during year 2 (N=4) to increase adult vaccination rates.
- Pittsburgh Control/Maintenance Sites: Practices: Clinical practices were stratified by metropolitan area (e.g., Pittsburgh) and then randomized into the intervention or control arms within strata.
  Patients: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 6/1/2012 to 5/31/2013 (Tdap, PCV) and 8/1/2012 to 1/31/2013 (influenza), Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Year 1 RCCT study: Control sites were Pittsburgh practices who did not receive the 4 Pillars Practice Transformation Program intervention until Year 2 (N=8).
  Year 2 Pre-post study: Maintenance sites were Pittsburgh practices who were intervened upon in Year 1 but who did not actively participate in continued engagement of the 4 Pillars Program for raising adult vaccination rates during Year 2 (N=6).
- Houston Intervention Sites: Practices: Clinical practices were stratified by metropolitan area (e.g., Houston) and then randomized into the intervention or control arms within strata.
  Patients: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 6/1/2012 to 5/31/2013 (Tdap, PCV) and 8/1/2012 to 1/31/2013 (influenza), Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Year 1 RCCT study: Intervention sites were Houston practices who actively utilized the 4 Pillars Practice Transformation Program during Year 1 to promote increases in adult vaccination rates (N=3).
  Year 2 Pre-post study: Year 2 Houston practices were control sites from Year 1 (N=3) who now were actively engaged in the intervention to increase adult vaccination rates.
- Houston Control/Maintenance Sites: Practices: Clinical practices were stratified by metropolitan area (e.g., Houston) and then randomized into the intervention or control arms within strata.
  Patients: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 6/1/2012 to 5/31/2013 (Tdap, PCV) and 8/1/2012 to 1/31/2013 (influenza), Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Year 1 RCCT study: Control sites were Houston practices who did not receive the 4 Pillars Practice Transformation Program intervention until Year 2 (N=3).
  Year 2 Pre-post study: Maintenance sites were Houston practices who were intervened upon in Year 1 but who did not actively participate in continued engagement of the 4 Pillars Program for raising adult vaccination rates during Year 2 (N=3).
Period: Year 1 RCCT Study
Arm/Group | Pittsburgh Intervention Sites | Pittsburgh Control/Maintenance Sites | Houston Intervention Sites | Houston Control/Maintenance Sites
Started | 13186; 10 clinical practices | 17185; 8 clinical practices | 19274; 3 clinical practices | 20904; 3 clinical practices
Completed | 13186; 10 clinical practices | 17185; 8 clinical practices | 19274; 3 clinical practices | 20904; 3 clinical practices
Not Completed | 0; 0 clinical practices | 0; 0 clinical practices | 0; 0 clinical practices | 0; 0 clinical practices
Period: Year 2 Pre-post Study
Arm/Group | Pittsburgh Intervention Sites | Pittsburgh Control/Maintenance Sites | Houston Intervention Sites | Houston Control/Maintenance Sites
Started | 22324; 12 clinical practices (Reflects: control sites from Year 1 (N=8) and Year 1 Intervention sites who continued in Y2 (N=4)) | 8047; 6 clinical practices (Reflects: the six Year 1 Intervention sites who chose not to actively engage Year 2) | 20904; 3 clinical practices (Reflects: Year 1 Control sites who became active in the intervention during Year 2) | 19274; 3 clinical practices (Reflects: Year 1 Intervention sites who chose not to actively engage Year 2)
Completed | 22324; 12 clinical practices | 8047; 6 clinical practices | 20904; 3 clinical practices | 19274; 3 clinical practices
Not Completed | 0; 0 clinical practices | 0; 0 clinical practices | 0; 0 clinical practices | 0; 0 clinical practices

BASELINE CHARACTERISTICS:
Population: Information provided for baseline demographics comes from the Tdap citation: Nowalk MP, Lin CJ, Pavlik VN, et al. Using the 4 Pillars™ Practice Transformation Program to increase adult Tdap immunization in a randomized controlled cluster trial. Vaccine. 2016 Sep 22;34(41):5026-33. Epub 2016 Aug 26. PubMed ID: 27576073
Units Other Than Participants: clinical practices
Groups:
- Pittsburgh Intervention: Practices: Represents 10 clinical practices engaged in active intervention in Year 1.
  Patients: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 6/1/2012 to 5/31/2013 (Tdap, pneumococcal) and 8/1/2012 to 1/31/2013 (influenza), Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 (Tdao, pneumococcal) and 8/1/2013 to 1/31/2014 (influenza) and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015 (Tdap, pneumococcal) and 8/1/2014 to 1/31/2015 (influenza).
- Pittsburgh Control/Maintenance: Practices: Represents 8 clinical practices who were control practices in Year 1 and who received the intervention in Year 2.
  Patients: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 6/1/2012 to 5/31/2013 (Tdap, pneumococcal) and 8/1/2012 to 1/31/2013 (influenza), Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 (Tdao, pneumococcal) and 8/1/2013 to 1/31/2014 (influenza) and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015 (Tdap, pneumococcal) and 8/1/2014 to 1/31/2015 (influenza).
- Houston Intervention: Practices: Represents 3 clinical practices engaged in active intervention in Year 1.
  Patients: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 6/1/2012 to 5/31/2013 (Tdap, pneumococcal) and 8/1/2012 to 1/31/2013 (influenza), Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 (Tdao, pneumococcal) and 8/1/2013 to 1/31/2014 (influenza) and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015 (Tdap, pneumococcal) and 8/1/2014 to 1/31/2015 (influenza).
- Houston Control/Maintenance: Practices: Represents 3 clinical practices who were control practices in Year 1 and who received the intervention in Year 2.
  Patients: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 6/1/2012 to 5/31/2013 (Tdap, pneumococcal) and 8/1/2012 to 1/31/2013 (influenza), Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 (Tdao, pneumococcal) and 8/1/2013 to 1/31/2014 (influenza) and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015 (Tdap, pneumococcal) and 8/1/2014 to 1/31/2015 (influenza).
- Total: Total of all reporting groups
Arm/Group | Pittsburgh Intervention | Pittsburgh Control/Maintenance | Houston Intervention | Houston Control/Maintenance | Total
Number analyzed (Participants) | 13,186 | 17,185 | 19,274 | 20,904 | 70549
Number analyzed (clinical practices) | 10 | 8 | 3 | 3 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (16.7) | 57.8 (16.6) | 51.0 (13.0) | 53.0 (13.0) | 55.1 (15.3)
Sex/Gender, Customized [Number; unit: percentage of participants]
  % Female Sex | 56.7 | 57.8 | 72.0 | 71.0 | 65.5
Race/Ethnicity, Customized [Number; unit: percentage of participants]
  % Caucasians | 94.3 | 94.2 | 6.0 | 7.0 | 44.3

OUTCOME MEASURES:

1. Primary Outcome: Year 1 RCCT: Change From Baseline in the Percentage of Participants Who Were Vaccinated at the End of Year 1
Description: Outcome listed is total percentage point difference in vaccination rates from baseline to end of year 1
Time Frame: % vaccinated by 5/31/2014 (Tdap, Pneumococcal); % vaccinated by 1/31/2014 (Influenza)
Measure: Number; unit: percent change in vaccination rates
Groups:
- Year 1 RCCT Pittsburgh Intervention Sites - Tdap Vaccination: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 6/1/2012 to 5/31/2013, Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Intervention sites were Pittsburgh practices who actively utilized the 4 Pillars Practice Transformation Program during Year 1 to promote increases in adult Tdap vaccination (N=10).
- Year 1 RCCT Pittsburgh Control Sites - Tdap Vaccination: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 6/1/2012 to 5/31/2013, Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Control sites were Pittsburgh practices who did not receive the 4 Pillars Practice Transformation Program intervention until Year 2 (N=8).
- Year 1 RCCT Pittsburgh Intervention Sites - Pneumococcal Vacc: Adults >=65 years of age at baseline who were active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 6/1/2012 to 5/31/2013, Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Intervention sites were Pittsburgh practices who actively utilized the 4 Pillars Practice Transformation Program during Year 1 to promote increases in adult PPSV vaccination (N=10).
- Year 1 RCCT Pittsburgh Control Sites - Pneumococcal Vaccine: Adults >=65 years of age at baseline who were active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 6/1/2012 to 5/31/2013, Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Control sites were Pittsburgh practices who did not receive the 4 Pillars Practice Transformation Program intervention until Year 2 (N=8).
- Year 1 RCCT Pittsburgh Intervention Sites - Influenza Vaccine: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 8/1/2012 to 1/31/2013, Year 1 period (which was the randomized controlled cluster trial) was 8/1/2013 to 1/31/2014 and Year 2 (a pre-post study) was 8/1/2014 to 1/31/2015.
  Intervention sites were Pittsburgh practices who actively utilized the 4 Pillars Practice Transformation Program during Year 1 to promote increases in adult influenza vaccination (N=10).
- Year 1 RCCT Pittsburgh Control Sites - Influenza Vaccine: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 8/1/2012 to 1/31/2013, Year 1 period (which was the randomized controlled cluster trial) was 8/1/2013 to 1/31/2014 and Year 2 (a pre-post study) was 8/1/2014 to 1/31/2015.
  Control sites were Pittsburgh practices who did not receive the 4 Pillars Practice Transformation Program intervention until Year 2 (N=8).
- Year 1 RCCT Houston Intervention Sites - Tdap Vaccination: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 6/1/2012 to 5/31/2013, Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Intervention sites were Houston practices who actively utilized the 4 Pillars Practice Transformation Program during Year 1 to promote increases in adult Tdap vaccination (N=3).
- Year 1 RCCT Houston Control Sites - Tdap Vaccination: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 6/1/2012 to 5/31/2013, Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Control sites were Houston practices who did not receive the 4 Pillars Practice Transformation Program intervention until Year 2 (N=3).
- Year 1 RCCT Houston Intervention Sites - Pneumococcal Vaccine: Adults >=65 years of age at baseline who were active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 6/1/2012 to 5/31/2013, Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Intervention sites were Houston practices who actively utilized the 4 Pillars Practice Transformation Program during Year 1 to promote increases in adult PPSV vaccination (N=3).
- Year 1 RCCT Houston Control Sites - Pneumococcal Vaccine: Adults >=65 years of age at baseline who were active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 6/1/2012 to 5/31/2013, Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Control sites were Houston practices who did not receive the 4 Pillars Practice Transformation Program intervention until Year 2 (N=3).
- Year 1 RCCT Houston Intervention Sites - Influenza Vaccination: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 8/1/2012 to 1/31/2013, Year 1 period (which was the randomized controlled cluster trial) was 8/1/2013 to 1/31/2014 and Year 2 (a pre-post study) was 8/1/2014 to 1/31/2015.
  Intervention sites were Houston practices who actively utilized the 4 Pillars Practice Transformation Program during Year 1 to promote increases in adult influenza vaccination (N=3).
- Year 1 RCCT Houston Control Sites - Influenza Vaccination: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Baseline period was 8/1/2012 to 1/31/2013, Year 1 period (which was the randomized controlled cluster trial) was 8/1/2013 to 1/31/2014 and Year 2 (a pre-post study) was 8/1/2014 to 1/31/2015.
  Control sites were Houston practices who did not receive the 4 Pillars Practice Transformation Program intervention until Year 2 (N=3).
Arm/Group | Year 1 RCCT Pittsburgh Intervention Sites - Tdap Vaccination | Year 1 RCCT Pittsburgh Control Sites - Tdap Vaccination | Year 1 RCCT Pittsburgh Intervention Sites - Pneumococcal Vacc | Year 1 RCCT Pittsburgh Control Sites - Pneumococcal Vaccine | Year 1 RCCT Pittsburgh Intervention Sites - Influenza Vaccine | Year 1 RCCT Pittsburgh Control Sites - Influenza Vaccine | Year 1 RCCT Houston Intervention Sites - Tdap Vaccination | Year 1 RCCT Houston Control Sites - Tdap Vaccination | Year 1 RCCT Houston Intervention Sites - Pneumococcal Vaccine | Year 1 RCCT Houston Control Sites - Pneumococcal Vaccine | Year 1 RCCT Houston Intervention Sites - Influenza Vaccination | Year 1 RCCT Houston Control Sites - Influenza Vaccination
Number analyzed (Participants) | 13,186 | 17,185 | 6,095 | 6,223 | 13,186 | 17,185 | 19,274 | 20,904 | 3,010 | 2,779 | 19,274 | 20,904
percent change in vaccination rates | 7.7 | 6.4 | 6.5 | 6.6 | 5.0 | 6.5 | 9.9 | 7.6 | 8.7 | 6.5 | 2.7 | 5.2
Statistical Analysis 1: Comparison: Year 1 RCCT Pittsburgh Intervention Sites - Tdap Vaccination vs Year 1 RCCT Pittsburgh Control Sites - Tdap Vaccination vs Year 1 RCCT Pittsburgh Intervention Sites - Pneumococcal Vacc vs Year 1 RCCT Pittsburgh Control Sites - Pneumococcal Vaccine vs Year 1 RCCT Houston Intervention Sites - Tdap Vaccination vs Year 1 RCCT Houston Control Sites - Tdap Vaccination vs Year 1 RCCT Houston Intervention Sites - Pneumococcal Vaccine vs Year 1 RCCT Houston Control Sites - Pneumococcal Vaccine; Test type: Superiority or Other; p = 0.05, Chi-squared; Chi-square tests for comparisons between-arm changes in vaccination rates between Baseline and Year 1 for RCCT study period
Statistical Analysis 2: Comparison: Year 1 RCCT Pittsburgh Intervention Sites - Influenza Vaccine vs Year 1 RCCT Pittsburgh Control Sites - Influenza Vaccine vs Year 1 RCCT Houston Intervention Sites - Influenza Vaccination vs Year 1 RCCT Houston Control Sites - Influenza Vaccination; Test type: Superiority or Other; p = 0.05, Cochran-Armitage trend test — Cochran-Armitage trend tests for percentage point difference between Baseline and Year 1 for RCCT study period

2. Secondary Outcome: Year 2 Pre-post Study: Change From Year 1 in the Percentage of Participants Who Were Vaccinated at the End of Year 2
Description: Outcome listed is total percentage point difference in vaccination rates from end of year 1 to end of year 2
Time Frame: % vaccinated by 1/31/2015
Measure: Number; unit: percent change in vaccination rates
Groups:
- Year 2 Pre-post Study Pittsburgh Intervention Sites - Tdap: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Year 2 Pittsburgh practices were control sites from Year 1 (N=8) who now were actively engaged in the intervention and Year 1 sites who continued active use of the intervention during year 2 (N=4) to increase adult Tdap vaccination rates.
- Year 2 Pre-post Study Pittsburgh Maintenance Sites - Tdap: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Maintenance sites were Pittsburgh practices who were intervened upon in Year 1 but who did not actively participate in continued engagement of the 4 Pillars Program for raising adult Tdap vaccination rates during Year 2 (N=6).
- Year 2 Pre-post Study Pittsburgh Intervention Sites - PPSV: Adults >=65 years of age at baseline who were active patients of 25 diverse practices who were seen >=1 time each year. Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Year 2 Pittsburgh practices were control sites from Year 1 (N=8) who now were actively engaged in the intervention and Year 1 sites who continued active use of the intervention during year 2 (N=4) to increase adult pneumococcal vaccination rates.
- Year 2 Pre-post Study Pittsburgh Maintenance Sites - PPSV: Adults >=65 years of age at baseline who were active patients of 25 diverse practices who were seen >=1 time each year. Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Maintenance sites were Pittsburgh practices who were intervened upon in Year 1 but who did not actively participate in continued engagement of the 4 Pillars Program for raising adult pneumococcal vaccination rates during Year 2 (N=6).
- Year 2 Pre-post Study Pittsburgh Intervention Sites-Influenza: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Year 1 period (which was the randomized controlled cluster trial) was 8/1/2013 to 1/31/2014 and Year 2 (a pre-post study) was 8/1/2014 to 1/31/2015.
  Year 2 Pittsburgh practices were control sites from Year 1 (N=8) who now were actively engaged in the intervention and Year 1 sites who continued active use of the intervention during year 2 (N=4) to increase adult influenza vaccination rates.
- Year 2 Pre-post Study Pittsburgh Maintenance Sites - Influenza: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Year 1 period (which was the randomized controlled cluster trial) was 8/1/2013 to 1/31/2014 and Year 2 (a pre-post study) was 8/1/2014 to 1/31/2015.
  Maintenance sites were Pittsburgh practices who were intervened upon in Year 1 but who did not actively participate in continued engagement of the 4 Pillars Program for raising adult influenza vaccination rates during Year 2 (N=6).
- Year 2 Pre-post Study Houston Intervention Sites - Tdap: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Year 2 Houston practices were control sites from Year 1 (N=3) who now were actively engaged in the intervention to increase adult Tdap vaccination rates.
- Year 2 Pre-post Study Houston Maintenance Sites - Tdap: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Maintenance sites were Houston practices who were intervened upon in Year 1 but who did not actively participate in continued engagement of the 4 Pillars Program for raising adult Tdap vaccination rates during Year 2 (N=3).
- Year 2 Pre-post Study Houston Intervention Sites - PPSV: Adults >=65 years of age at baseline who were active patients of 25 diverse practices who were seen >=1 time each year. Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Year 2 Houston practices were control sites from Year 1 (N=3) who now were actively engaged in the intervention to raise adult pneumococcal vaccination rates.
- Year 2 Pre-post Study Houston Maintenance Sites - PPSV: Adults >=65 years of age at baseline who were active patients of 25 diverse practices who were seen >=1 time each year. Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  Maintenance sites were Houston practices who were intervened upon in Year 1 but who did not actively participate in continued engagement of the 4 Pillars Program for raising adult pneumococcal vaccination rates during Year 2 (N=3).
- Year 2 Pre-post Study Houston Intervention Sites - Influenza: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Year 1 period (which was the randomized controlled cluster trial) was 8/1/2013 to 1/31/2014 and Year 2 (a pre-post study) was 8/1/2014 to 1/31/2015.
  Year 2 Houston practices were control sites from Year 1 (N=3) who now were actively engaged in the intervention to increase adult influenza vaccination rates.
- Year 2 Pre-post Study Houston Maintenance Sites - Influenza: Adults > 18 years of age who are active patients of 25 diverse practices who were seen >=1 time each year. Year 1 period (which was the randomized controlled cluster trial) was 8/1/2013 to 1/31/2014 and Year 2 (a pre-post study) was 8/1/2014 to 1/31/2015.
  Maintenance sites were Houston practices who were intervened upon in Year 1 but who did not actively participate in continued engagement of the 4 Pillars Program for raising adult influenza vaccination rates during Year 2 (N=3).
Arm/Group | Year 2 Pre-post Study Pittsburgh Intervention Sites - Tdap | Year 2 Pre-post Study Pittsburgh Maintenance Sites - Tdap | Year 2 Pre-post Study Pittsburgh Intervention Sites - PPSV | Year 2 Pre-post Study Pittsburgh Maintenance Sites - PPSV | Year 2 Pre-post Study Pittsburgh Intervention Sites-Influenza | Year 2 Pre-post Study Pittsburgh Maintenance Sites - Influenza | Year 2 Pre-post Study Houston Intervention Sites - Tdap | Year 2 Pre-post Study Houston Maintenance Sites - Tdap | Year 2 Pre-post Study Houston Intervention Sites - PPSV | Year 2 Pre-post Study Houston Maintenance Sites - PPSV | Year 2 Pre-post Study Houston Intervention Sites - Influenza | Year 2 Pre-post Study Houston Maintenance Sites - Influenza
Number analyzed (Participants) | 22,324 | 8,047 | 8,326 | 3,992 | 22,324 | 8,047 | 20,904 | 19,274 | 2,779 | 3,010 | 20,904 | 19,274
percent change in vaccination rates | 6.2 | 2.2 | 5.2 | 2.4 | 1.44 | 1.4 | 6.2 | 4.1 | 4.6 | 6.5 | 3.6 | 1.7
Statistical Analysis 1: Comparison: Year 2 Pre-post Study Pittsburgh Intervention Sites - Tdap vs Year 2 Pre-post Study Pittsburgh Maintenance Sites - Tdap vs Year 2 Pre-post Study Pittsburgh Intervention Sites - PPSV vs Year 2 Pre-post Study Pittsburgh Maintenance Sites - PPSV vs Year 2 Pre-post Study Houston Intervention Sites - Tdap vs Year 2 Pre-post Study Houston Maintenance Sites - Tdap vs Year 2 Pre-post Study Houston Intervention Sites - PPSV vs Year 2 Pre-post Study Houston Maintenance Sites - PPSV; Test type: Superiority or Other; p = 0.05, Chi-squared; Chi-square tests for comparisons between-arm changes in vaccination rates between pre and post intervention for Pre-post study period
Statistical Analysis 2: Comparison: Year 2 Pre-post Study Pittsburgh Intervention Sites-Influenza vs Year 2 Pre-post Study Pittsburgh Maintenance Sites - Influenza vs Year 2 Pre-post Study Houston Intervention Sites - Influenza vs Year 2 Pre-post Study Houston Maintenance Sites - Influenza; Test type: Superiority or Other; p = 0.05, Cochran-Armitage trend test — Cochran-Armitage trend tests for difference between pre and post changes in vaccination rates for Pre-Post study period

ADVERSE EVENTS:
Time Frame: 3 years (Baseline, Year 1, Year 2)
Description: For the Tdap and Pneumococcal cohorts: Baseline period was 6/1/2012 to 5/31/2013, Year 1 period (which was the randomized controlled cluster trial) was 6/1/2013 to 5/31/2014 and Year 2 (a pre-post study) was 6/1/2014 to 1/31/2015.
  For the Influenza cohort: Baseline period was 8/1/2012 to 1/31/2013, Year 1 period (which was the randomized controlled cluster trial) was 8/1/2013 to 1/31/2014 and Year 2 (a pre-post study) was 8/1/2014 to 1/31/2015.
Arm/Group | Year 1 RCCT Pittsburgh Intervention Sites - Tdap Vaccination | Year 1 RCCT Pittsburgh Control Sites - Tdap Vaccination | Year 1 RCCT Pittsburgh Intervention Sites - Pneumococcal Vacc | Year 1 RCCT Pittsburgh Control Sites - Pneumococcal Vaccine | Year 1 RCCT Pittsburgh Intervention Sites - Influenza Vaccine | Year 1 RCCT Pittsburgh Control Sites - Influenza Vaccine | Year 1 RCCT Houston Intervention Sites - Tdap Vaccination | Year 1 RCCT Houston Control Sites - Tdap Vaccination | Year 1 RCCT Houston Intervention Sites - Pneumococcal Vaccine | Year 1 RCCT Houston Control Sites - Pneumococcal Vaccine | Year 1 RCCT Houston Intervention Sites - Influenza Vaccination | Year 1 RCCT Houston Control Sites - Influenza Vaccination
All-Cause Mortality (participants affected / at risk) | 0/13186 | 0/17185 | 0/6095 | 0/6223 | 0/13186 | 0/17185 | 0/19274 | 0/20904 | 0/3010 | 0/2779 | 0/19274 | 0/20904
Serious Adverse Events (participants affected / at risk) | 0/13186 | 0/17185 | 0/6095 | 0/6223 | 0/13186 | 0/17185 | 0/19274 | 0/20904 | 0/3010 | 0/2779 | 0/19274 | 0/20904
Other Adverse Events (participants affected / at risk) | 0/13186 | 0/17185 | 0/6095 | 0/6223 | 0/13186 | 0/17185 | 0/19274 | 0/20904 | 0/3010 | 0/2779 | 0/19274 | 0/20904

LIMITATIONS AND CAVEATS:
The limitations of this study included late delivery of influenza vaccine in Year 1 in the Pittsburgh sites, delay of EMR data for reporting study progress to sites (all vaccines) and vaccine increases in control arm (Tdap and PPSV) during Year 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No